CLINICAL TRIAL: NCT02274519
Title: Novel Support Options in Autologous Stem Cell Transplant for Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Nandita Khera, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-007210
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Multiple Myeloma; Plasma Cell Disorder
Keywords: multiple myeloma; plasma cell disorder; autologous stem cell transplant
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Tai Ji; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tai Chi (Experimental): Group randomized to participate in Tai Chi intervention
  Interventions: Other: Tai Chi
- Educational (Active Comparator): Group randomized to participate in educational intervention
  Interventions: Other: Education

INTERVENTIONS:
Other: Tai Chi — Arm 1
  Arms: Tai Chi
Other: Education — Arm 2
  Arms: Educational

SUMMARY:
Does Tai Chi Easy (TCEasy), a simple and repetitive form of exercise that consists of movements with meditation, improve quality of life in those afflicted with multiple myeloma undergoing autologous stem cell transplantation?

DETAILED DESCRIPTION:
All patients with Multiple Myeloma seen at Mayo Clinic Arizona who are undergoing evaluation for autologous stem cell transplant will be identified for potential candidacy by BMT transplant coordinator staff and referred to CRC study staff for final screen of candidacy over a period of 12 months. If eligible, ≤ 30 days prior to transplant CRC study staff will meet with patient for consent and undergo 1:1 randomization to Tai Chi versus educational control arm (N: 70). No earlier than 7 days prior to transplant all patients will attend a 1 hour session consisting of Tai Chi techniques or receive educational materials depending on the patients prior randomization and will start their intervention, subject diary and support materials will be provided. Patients will be asked to perform 30 minutes of intervention daily (Tai Chi versus educational control) and document minutes and quality of practice in their subject diary. On day 1 of autologous stem cell transplant CRC staff will administer the baseline questionnaires (NIH PROMIS Short form questionnaires for pain, depression, anxiety, social isolation, and sleep). Patients will continue their intervention (Tai chi versus educational control) daily throughout autologous stem cell transplant and record intervention fidelity in patient diary. On day 14 of transplant the NIH PROMIS questionnaires, perceived benefit questionnaire, and the meditative movement inventory for the Tai chi group only will be collected. Data collection for secondary outcomes including time to engraftment, incidence of febrile neutropenia, days of hospitalization, etc will be also gathered. Patients will continue intervention through transplant day 30 (+/- 5 days) at which time, CRC staff will collect subject diary, administer NIH PROMIS questionnaires, and a perceived benefit questionnaire. Adherence reminders will be executed once per week by CRC staff from date of initiation of intervention to completion of study.

The intervention to be tested, TCEasy, is a standardized protocol that was developed by Dr. Roger Jahnke and has been used in several prior studies including a recently completed NIH/NCCAM-funded randomized controlled trial (RCT) with breast cancer survivors (U01 AT002706-03: PI Linda Larkey, PhD, Arizona State University, primary outcome paper currently under review). Participants will be given a written instruction manual for the Tai Chi exercises to refer to after training has been administered.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Multiple myeloma > 18 years of age or greater
* English speaking
* General proficiency to read and write in English
* Able to attend training session per study protocol
* ECOG performance status 0-1

Exclusion Criteria:

* Currently performs Tai Chi, Qi Gong, or Yoga at least once weekly or more
* Syncopal event in prior 60 days
* Current Grade 3 or > neuropathy
* Concurrent major depressive disorder or anxiety disorder (DSMIV)
* Chronic Dizziness and/or vestibular disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-02; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Quality of life | 30 days
  Quality of life measures including pain, depression, anxiety, social isolation, and sleep utilizing NIH promis SF series

SECONDARY OUTCOMES:
Time to engraftment | 15 days
Rate of febrile neutropenia | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Nandita Khera, MD, MPH, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials